CLINICAL TRIAL: NCT06647758
Title: Association Between Remote Post-operative Anemia and Mortality in Patients Undergoing Valvular Heart Surgery
Brief Title: Association Between Post-operative Anemia and Mortality After Valvular Heart Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2024-0674
Record Dates: First submitted 2024-10-13; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Patients Undergoing Valvular Heart Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- preoperative anemia-postoperative anemia
- preopertive anemia-postoperitve non-anemia
- preoperative non-anemia-postoperative anemia
- preopeartive non-anemia-postopertive non-anemia

SUMMARY:
The investigators aimed to evaluate whether postoperative anemia can predict 1-year mortality after valvular heart surgery independent of preoperative anemia. Patients who underwent valvular heart surgery were divided into four groups according to whether or not they had preoperative and postoperative anemia. Postoperative one-year mortality, as well as overall mortality and a composite of death and heart failure requiring hospitalization, was investigated according to the groups, adjusted by confounders.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent valvular heart surgery between January 2016 and July 2023 at Severance Cardiovascular Hospital of Yonsei University Health System.

Exclusion Criteria:

* patients who underwent only pulmonary valve surgery
* those with missing hemoglobin values at 2months after the surgery, due to loss of follow up or death.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: tertiary care hospital
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-07-21 (Estimated); Study Completion 2025-07-21 (Estimated)

PRIMARY OUTCOMES:
postoperative 1-year mortality | One year after valvular heart surgery
  The investigators assessed all-cause mortality during one year after valvular heart surgery and evaluated its association with preoperative and postoperative anemic status.

SECONDARY OUTCOMES:
overall mortality | postopeartive one-year
  The investigators assessed overall mortality during the follow-up period and a composite of death and congestive heart failure (CHF) requiring rehospitalization during the postoperative one-year and evaluated their associations with preoperative and postoperative anemic status.
composite of death and congestive heart failure (CHF) requiring rehospitalization | postopeartive one-year
  The investigators assessed overall mortality during the follow-up period and a composite of death and congestive heart failure (CHF) requiring rehospitalization during the postoperative one-year and evaluated their associations with preoperative and postoperative anemic status.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine and Anesthesia, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No